CLINICAL TRIAL: NCT06274060
Title: Optimizing PrEP Implementation and Effectiveness Among Women at High Risk for HIV Acquisition in South Africa: Phase 2b
Brief Title: Project Phakama: Testing Support Strategies to Empower Young Women on PrEP in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: TB HIV Care (Other); Unity Health Toronto (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 135399; R01MH121161 (NIH); IRB00012628 (Other: JHSPH IRB)
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Pre-exposure Prophylaxis; HIV Infections
Keywords: PrEP; HIV prevention; Adolescent girls and young women; Female sex workers; South Africa
MeSH Terms: conditions — HIV Infections | interventions — Case Management

STUDY DESIGN:
Intervention Model Description: This fractional factorial design includes four strategies resulting in 16 trial arms/conditions. The design compares results in arms with and without each of the strategies, but is not fully powered to test every combination of strategies.Thus, each strategy will be received by half of the participants, though the combinations of strategies will vary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Standard of care (No Intervention): The TB HIV Care programme standard of care includes full-time peer educators employed by the programme to engage women, layered PrEP promotion across prevention programmes, and "refer a friend" strategies, information, education and communication (IEC) materials, service user testimonials, risk reduction posters to better align young women's perception of risk, working after hours/weekends to reach young women, working with school governing bodies, and door-to-door outreach.
- Case management (Experimental): Participants will receive case management layered on existing standard of care.
  Interventions: Behavioral: Case management
- Food vouchers (Experimental): Participants will receive food vouchers layered on existing standard of care.
  Interventions: Behavioral: Food vouchers
- PrEP support buddy (Experimental): Participants will receive the PrEP support buddy intervention layered on existing standard of care.
  Interventions: Behavioral: PrEP support buddy
- Community-based PrEP pickup points (Experimental): Participants will receive the community-based PrEP pickup point intervention layered on existing standard of care.
  Interventions: Behavioral: Community-based PrEP pickup points
- PrEP support buddy + Community-based PrEP pickup points (Experimental): Participants in this arm will receive both the PrEP support buddy and community-based PrEP pickup point interventions in combination.
  Interventions: Behavioral: PrEP support buddy; Behavioral: Community-based PrEP pickup points
- Food vouchers + Community-based PrEP pickup points (Experimental): Participants in this arm will receive both the food voucher and community-based PrEP pickup point interventions in combination.
  Interventions: Behavioral: Food vouchers; Behavioral: Community-based PrEP pickup points
- Food vouchers + PrEP support buddy (Experimental): Participants in this arm will receive both the food voucher and PrEP support buddy interventions in combination.
  Interventions: Behavioral: Food vouchers; Behavioral: PrEP support buddy
- Case management + Community-based PrEP pickup points (Experimental): Participants in this arm will receive both the case management and community-based PrEP pickup point interventions in combination.
  Interventions: Behavioral: Case management; Behavioral: Community-based PrEP pickup points
- Case management + PrEP support buddy (Experimental): Participants in this arm will receive both the case management and PrEP support buddy interventions in combination.
  Interventions: Behavioral: Case management; Behavioral: PrEP support buddy
- Case management + Food vouchers (Experimental): Participants in this arm will receive both the case management and food voucher interventions in combination.
  Interventions: Behavioral: Case management; Behavioral: Food vouchers
- Food voucher + PrEP support buddy + Community-based PrEP pickup points (Experimental): Participants in this arm will receive the food voucher, PrEP support buddy, and community-based PrEP pickup point interventions in combination.
  Interventions: Behavioral: Food vouchers; Behavioral: PrEP support buddy; Behavioral: Community-based PrEP pickup points
- Case management + PrEP support buddy + Community-based PrEP pickup points (Experimental): Participants in this arm will receive the case management, PrEP support buddy, and community-based PrEP pickup point interventions in combination.
  Interventions: Behavioral: Case management; Behavioral: PrEP support buddy; Behavioral: Community-based PrEP pickup points
- Case management + Food vouchers + Community-based PrEP pickup points (Experimental): Participants in this arm will receive the case management, food vouchers, and community-based PrEP pickup point interventions in combination.
  Interventions: Behavioral: Case management; Behavioral: Food vouchers; Behavioral: Community-based PrEP pickup points
- Case management + Food vouchers + PrEP support buddy (Experimental): Participants in this arm will receive the case management, food vouchers, and PrEP support buddy interventions in combination.
  Interventions: Behavioral: Case management; Behavioral: Food vouchers; Behavioral: PrEP support buddy
- Case management + Food vouchers + PrEP support buddy + Community-based PrEP pickup points (Experimental): Participants in this arm will receive the case management, food vouchers, PrEP support buddy, and community-based PrEP pickup point interventions in combination.
  Interventions: Behavioral: Case management; Behavioral: Food vouchers; Behavioral: PrEP support buddy; Behavioral: Community-based PrEP pickup points

INTERVENTIONS:
Behavioral: Case management — Participants will receive case management delivered by a peer with PrEP experience/success for seven months, with the goal of improving self-efficacy to take PrEP. The intention of this intervention is to help participants to develop individualized strategies to address and overcome barriers to PrEP use, as well as develop disclosure strategies. This strategy includes weekly face-to-face support with the case manager for the first month of the trial, followed by monthly face-to-face support for the remainder of the trial follow up period. The strategy will also include client-initiated on-demand phone consultation with the case manager and mental health/substance use screening and referrals. Participants randomized to this strategy may also opt into daily timed PrEP pill-taking reminders via short message service (SMS).
  Arms: Case management; Case management + Community-based PrEP pickup points; Case management + Food vouchers; Case management + Food vouchers + Community-based PrEP pickup points; Case management + Food vouchers + PrEP support buddy; Case management + Food vouchers + PrEP support buddy + Community-based PrEP pickup points; Case management + PrEP support buddy; Case management + PrEP support buddy + Community-based PrEP pickup points
Behavioral: Food vouchers — Participants will be given food vouchers with a value of 200 South African Rand at the time of PrEP initiation and at 1- and 4-month standard of care visits at which clinical checkups and PrEP refills are provided. The goal of these vouchers is to improve participants' capacity to persist on PrEP. While PrEP can be taken without food, some experience increased side effects or prefer to take pills with food, making adherence difficult if they cannot afford food at times.
  Arms: Case management + Food vouchers; Case management + Food vouchers + Community-based PrEP pickup points; Case management + Food vouchers + PrEP support buddy; Case management + Food vouchers + PrEP support buddy + Community-based PrEP pickup points; Food voucher + PrEP support buddy + Community-based PrEP pickup points; Food vouchers; Food vouchers + Community-based PrEP pickup points; Food vouchers + PrEP support buddy
Behavioral: PrEP support buddy — Participants will identify a person in their network (such as a friend, partner, parent) that they wish to support them in their PrEP usage, with the goal of improving participants' motivation and self-efficacy to persist on PrEP and providing social support to facilitate ongoing PrEP use. Support buddies selected by FSW and AGYW randomized to this intervention will receive a one-time training session on PrEP and support strategies as well as informational materials and text reminders to assist them in providing ongoing PrEP support.
  Arms: Case management + Food vouchers + PrEP support buddy; Case management + Food vouchers + PrEP support buddy + Community-based PrEP pickup points; Case management + PrEP support buddy; Case management + PrEP support buddy + Community-based PrEP pickup points; Food voucher + PrEP support buddy + Community-based PrEP pickup points; Food vouchers + PrEP support buddy; PrEP support buddy; PrEP support buddy + Community-based PrEP pickup points
Behavioral: Community-based PrEP pickup points — Participants will be able to pick up PrEP from alternative pick-up points within the community that are convenient for them, with the goal of making PrEP more accessible to participants. Ten pickup points will be established at existing Hubs of Hope throughout the subdistricts served by the TB HIV Care programme. Hubs of Hope are based in the War Rooms within subdistricts, where the TB HIV Care programme operates, and serve as meeting places for service users to receive support searching for jobs, completing online courses, and other personal development activities to support a multi-sectoral approach to health. A TB HIV Care ambassador is based at each Hub of Hope to coordinate activities and provide support to service users. Participants who choose to use pick-up points will have the option of either completing an HIV self-test or testing with the on-site TB HIV Care staff to confirm HIV-negative status prior to receipt of PrEP refills.
  Arms: Case management + Community-based PrEP pickup points; Case management + Food vouchers + Community-based PrEP pickup points; Case management + Food vouchers + PrEP support buddy + Community-based PrEP pickup points; Case management + PrEP support buddy + Community-based PrEP pickup points; Community-based PrEP pickup points; Food voucher + PrEP support buddy + Community-based PrEP pickup points; Food vouchers + Community-based PrEP pickup points; PrEP support buddy + Community-based PrEP pickup points

SUMMARY:
The goal of this trial is to understand which strategies work best to support pre-exposure prophylaxis (PrEP) use among female sex workers (FSW) and adolescent girls and youth women (AGYW) in uMgungundlovu, KwaZulu-Natal, South Africa. Participants will be randomly assigned to receive a combination of up to four support strategies encourage the participants in continuing to use PrEP. The four strategies being tested are: case management, food vouchers, peer support buddies, and community-based PrEP pick-up points. The intention of this trial is to determine which PrEP support strategy or bundle(s) of strategies best promote(s) long-term PrEP use, so that these services can be scaled up to other districts in South Africa.

DETAILED DESCRIPTION:
The overall aim of this trial is to investigate which PrEP support strategies most effectively and efficiently optimize(s) PrEP persistence among female sex workers (FSW) and adolescent girls and youth women (AGYW) in South Africa. The trial will be implemented by TB HIV Care, a South African non-profit organization that provides direct HIV service delivery to FSW and AGYW across 10 districts in South Africa. The investigators plan to individually randomize 304 FSW and AGYW at the TB HIV Care site in uMgungundlovu, KwaZulu-Natal, to a fractional factorial trial, randomizing combinations of four separate strategies to support PrEP continuation. As fthe strategies are being tested, this results in 16 different intervention/study conditions, with one condition serving as a control where FSW and AGYW will receive the standard of care and no additional PrEP support. The other 15 conditions will be a combination of the standard of care alongside different PrEP delivery and support strategies implemented by TB HIV Care: case management, food vouchers, peer support buddies, and PrEP pick-up points. The intention of this trial is to determine which PrEP support strategy or bundle(s) of strategies best promote(s) long-term PrEP use and persistence, so that these services can be scaled up to other TB HIV Care sites. By utilizing the fractional factorial design in alignment the multiphase optimization strategy framework (MOST) the trial is feasible to conduct even with 16 arms, as the design compares results in arms with and without each of the strategies, but is not fully powered to test every combination of strategies.Thus, each strategy will be received by half of the participants, though the combinations of strategies will vary.

ELIGIBILITY:
Inclusion Criteria:

* Initiated PrEP within the past 48 hours by the TB HIV Care PrEP programme in uMgungundlovu through the female sex worker (FSW) or adolescent girls and young women (AGYW) PrEP programme teams

Exclusion Criteria:

* Not eligible for PrEP
* Currently on PrEP, but initiated onto PrEP more than 48 hours previously
* Under 16 years of age if AGYW OR under 18 years of age if FSW

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Identifies as a cisgender woman (assigned female sex at birth and currently identifies as a woman).
Enrollment: 304 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
PrEP persistence at 7 months after PrEP initiation | Month 7
  Proportion of trial participants who returned for their 7-month PrEP refill visit.
PrEP adherence at 7 months after PrEP initiation among all trial participants | Month 7
  The investigators will use dried blood spot (DBS) samples to measure PrEP adherence as an indicator of actual pill-taking. High PrEP adherence will be defined as taking 4 doses or more/week, measured as tenofovir-diphosphate (TFV-DP) ≥700 femtomoles per DBS sample. Among participants that do not return for DBS, the investigators will assume non-adherence and they will be included in this outcome.

SECONDARY OUTCOMES:
PrEP persistence at 1 month after PrEP initiation | Month 1
  Proportion of trial participants who returned for their 1-month PrEP refill visit.
PrEP persistence at 4 months after PrEP initiation | Month 4
  Proportion of trial participants who returned for their 4-month PrEP refill visit.
PrEP persistence at 13 months after PrEP initiation | Month 13
  Proportion of trial participants who returned for their 13-month PrEP refill visit.
PrEP adherence at 7 months after PrEP initiation among trial participants who provided dried blood spot samples | Month 7
  The investigators will use dried blood spot (DBS) samples to measure PrEP adherence as an indicator of actual pill-taking. High PrEP adherence will be defined as taking 4 doses or more/week, measured as tenofovir-diphosphate (TFV-DP) ≥700 femtomoles per DBS sample. Those who do not return at 7-months or do not provide a DBS sample will be excluded from this analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sheree Schwartz, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Harry Hausler, MD, PhD, MPH, Principal Investigator — TB HIV Care
Locations (1):
- TB HIV Care, Pietermaritzburg, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No